CLINICAL TRIAL: NCT01025778
Title: Clofarabine Based Remission Induction Followed by Haploidentical Stem Cell Transplantation in Children With Refractory Hematological Malignancies
Brief Title: Haploidentical Stem Cell Transplantation for Children With Therapy Resistant Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Jacek Toporski, MD, PhD, Head, Section of Pediatric Oncology/Hematology, Lund University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUS2009/1
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia
Keywords: Haploidentical hematopoietic stem cell transplantation; Graft versus host disease; Donor lymphocyte infusion; Graft versus leukemia effect; Immunological recovery; Bridge to transplant approach; Therapy resistant leukemia; Hematological malignancy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Graft vs Host Disease; Hematologic Neoplasms | interventions — Clofarabine; Remission Induction; Etoposide; Cyclophosphamide; Thiotepa; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remission induction and haplo-SCT (Experimental): Remission induction with Clofaranie, Etoposide and Cyclophosphamide combination followed by haplidentical stem cella transplantation if remission achieved.
  Interventions: Drug: Clofarabine for remission induction; Drug: Etoposide for remission induction; Drug: Cyclophosphamide for remission induction; Drug: Clofarabine in conditioning before transplantation; Drug: Thiotepa in conditioning before transplantation; Drug: Melfalan in conditioning before transplantation; Procedure: Haploidentical transplantation of T-cell depleted graft; Procedure: Donor lymphocyte infusion

INTERVENTIONS:
Drug: Clofarabine for remission induction
Drug: Etoposide for remission induction
Drug: Cyclophosphamide for remission induction
Drug: Clofarabine in conditioning before transplantation
Drug: Thiotepa in conditioning before transplantation
Drug: Melfalan in conditioning before transplantation
Procedure: Haploidentical transplantation of T-cell depleted graft
Procedure: Donor lymphocyte infusion

SUMMARY:
Despite substantial progress in the treatment pediatric acute leukemia a significant number of children will experience primary or secondary resistance to the treatment. In other words it will be not possible to achieve remission using standard chemotherapy (primary resistance) or the patients will develop chemotherapy resistant relapse (secondary resistance). Children failing to achieve remission or children relapsing after previous allogeneic stem cell transplantation have short life expectancy and palliative treatment still remains the most reasonable option as the escalation of conventional chemotherapy is not longer effective.

The role of Graft versus Leukemia effect was postulated as one of the mechanisms contributing to the leukemia control/eradication after transplantation of hematopoietic stem cells.

In this study the investigators combine intensified multiagent Clofarabine containing chemotherapy with post-induction treatment intensification using reduced intensity conditioning followed by haploidentical hematopoietic stem cell transplantation. Introducing a new drug to the treatment of resistant leukemia the investigators want to achieve a response which allows us to proceed to immediate haploidentical transplantation. Using a haploidentical donor the investigators can avoid time consuming search for an unrelated donor and perform the transplantation at the optimal time-point. Combating therapy resistant leukemia the investigators would like to evoke and utilize potential Graft-versus-Leukemia effect which is much more pronounced in the haploidentical setting, as it is well documented that allogeneic transplantation with a matched donor is not effective in resistant disease. The use of best KIR mismatch donor and post-transplant donor lymphocyte infusion will be implemented in order to develop/intensify graft versus leukemia effect.

ELIGIBILITY:
Inclusion Criteria:

Target population

1. Refractory acute lymphoblastic leukemia

   * Chemoresistant isolated or combined bone marrow relapse

     * Relapse after during/after conventional treatment
     * Relapse ≥6 months after allogeneic stem cell transplantation
   * Primary induction failure
   * Isolated extramedullary relapse after previous HSCT (>6 months)
2. Refractory acute myeloblastic leukemia including sAML

   * Chemoresistant relapse

     * Relapse after during/after conventional treatment
     * Relapse ≥6 months after allogeneic stem cell transplantation
   * Primary induction failure

Inclusion criteria to start induction treatment with multidrug regimen

1. Age ≥ 1 and ≤21 years
2. Patients with previous HCST ≥ 6 m
3. Provide signed written informed consent patients', and patients' parents /guardians

   * Older children should be capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent as well.
4. Cardiac output SF ≥25%
5. Have adequate renal and hepatic functions as indicated by the following laboratory values:

   * Calculated creatinine clearance ≥90 ml/min/1.73 m2
   * Serum bilirubin ≤1.5 X upper limit of normal (ULN)
   * Aspartate transaminase (AST)/alanine transaminase (ALT) ≤2.5 X ULN
   * Alkaline phosphatase ≤ 2.5 X ULN
6. Performance score of ≥70% (Lansky or Karnofsky)
7. A suitable haploidentical family member available for stem cell donation, > 18 years of age, fulfilling institutional criteria for blood and marrow donation.
8. Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Inclusion criteria to proceed to transplant after induction

1. Cardiac output SF ≥25%
2. Have adequate renal and hepatic functions as indicated by the following laboratory values:

   * Calculated creatinine clearance ≥90 ml/min/1.73 m2
   * Serum bilirubin ≤1.5 X upper limit of normal (ULN)
   * Aspartate transaminase (AST)/alanine transaminase (ALT) ≤2.5 X ULN
   * Alkaline phosphatase ≤ 2.5 X ULN
3. Performance score of ≥70% (Lansky or Karnofsky)
4. A suitable haploidentical family member available for stem cell donation, > 18 years of age, fulfilling institutional criteria for blood and marrow donation.
5. Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
6. Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
7. Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

1. Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
2. Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea.

   The patient must have recovered from all acute toxicities from any previous therapy.
3. Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
4. Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
5. Pregnant or lactating patients.
6. Any significant concurrent malignant disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Event free survival | 1 year from transplantation

SECONDARY OUTCOMES:
Evaluation of induction efficacy by response rate and the number of children proceeding to transplant | 3 months from induction start
Tolerance, safety and quality of life | 1 year from transplantation
Hematological and immunological recovery | 100 days fron tranplantation
Incidence of graft versus host disease | 100 days from transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Toporski, MD, PhD, Principal Investigator — Lund University Hospital
Locations (1):
- Lund University Hospital, Lund, Sweden

REFERENCES:
- [Background] Locatelli F, Testi AM, Bernardo ME, Rizzari C, Bertaina A, Merli P, Pession A, Giraldi E, Parasole R, Barberi W, Zecca M. Clofarabine, cyclophosphamide and etoposide as single-course re-induction therapy for children with refractory/multiple relapsed acute lymphoblastic leukaemia. Br J Haematol. 2009 Nov;147(3):371-8. doi: 10.1111/j.1365-2141.2009.07882.x. Epub 2009 Aug 29. PMID 19747360
- [Background] Hijiya N, Gaynon P, Barry E, Silverman L, Thomson B, Chu R, Cooper T, Kadota R, Rytting M, Steinherz P, Shen V, Jeha S, Abichandani R, Carroll WL. A multi-center phase I study of clofarabine, etoposide and cyclophosphamide in combination in pediatric patients with refractory or relapsed acute leukemia. Leukemia. 2009 Dec;23(12):2259-64. doi: 10.1038/leu.2009.185. Epub 2009 Sep 10. PMID 19741725
- [Background] Stern M, Ruggeri L, Mancusi A, Bernardo ME, de Angelis C, Bucher C, Locatelli F, Aversa F, Velardi A. Survival after T cell-depleted haploidentical stem cell transplantation is improved using the mother as donor. Blood. 2008 Oct 1;112(7):2990-5. doi: 10.1182/blood-2008-01-135285. Epub 2008 May 20. PMID 18492955
- [Background] Jeha S, Gaynon PS, Razzouk BI, Franklin J, Kadota R, Shen V, Luchtman-Jones L, Rytting M, Bomgaars LR, Rheingold S, Ritchey K, Albano E, Arceci RJ, Goldman S, Griffin T, Altman A, Gordon B, Steinherz L, Weitman S, Steinherz P. Phase II study of clofarabine in pediatric patients with refractory or relapsed acute lymphoblastic leukemia. J Clin Oncol. 2006 Apr 20;24(12):1917-23. doi: 10.1200/JCO.2005.03.8554. PMID 16622268
- [Result] Toporski J, Krol L, Dykes J, Hakansson Y, Pronk C, Turkiewicz D. The combination of clofarabine, etoposide, and cyclophosphamide shows limited efficacy as a bridge to transplant for children with refractory acute leukemia: results of a monitored prospective study. Pediatr Hematol Oncol. 2021 Apr;38(3):216-226. doi: 10.1080/08880018.2020.1838012. Epub 2020 Nov 5. PMID 33150834